CLINICAL TRIAL: NCT01519193
Title: Treatment of Aggressive Behavior and Post-Traumatic Stress Disorder in Former Street Children and Vulnerable Children in Burundi With Narrative Exposure Therapy for Violent Offenders
Brief Title: Treatment of Aggressive Behavior and Post-Traumatic Stress Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Konstanz (Other)
Responsible Party: Principal Investigator, Anselm Crombach, Principal Investigator, University of Konstanz
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: UKCR2011
Record Dates: First submitted 2011-12-01; First posted 2012-01-26 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Aggressive Behavior; Post-Traumatic Stress Disorder
Keywords: Aggressive Behavior; Appetitive Aggression; Post-Traumatic Stress Disorder
MeSH Terms: conditions — Aggression; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Narrative Exposure Therapy (Experimental)
  Interventions: Behavioral: Narrative Exposure Therapy for violent offenders (NETvo)
- No treatment control (No Intervention)

INTERVENTIONS:
Behavioral: Narrative Exposure Therapy for violent offenders (NETvo) — During NETvo the client, with the assistance of the therapist, constructs a chronological narrative of his whole life with a focus on exposure to traumatic stress and also on perpetrated violent acts. Empathic understanding, active listening, congruency and unconditional positive regard are key components of the therapist's behavior who asks in detail for emotions, cognitions, sensory information, and physiological reactions, linking them to an autobiographical context. Positive emotions and cognitions reported for violent acts are linked to the respective past. During four sessions the most important traumatic experiences and perpetrated violent acts are processed. In the fifth session plans and ideas for the future are developed to assist the children to reintegrate themselves into society.
  Arms: Narrative Exposure Therapy

SUMMARY:
Street children and children of vulnerable families in conflict or former conflict regions are often exposed to multiple traumatic events and situations in which they are forced to engage in violent behavior. The Narrative Exposure Therapy for violent offenders (NETvo) aims to reduce both PTSD symptoms and aggressive behavior. It helps the children to anchor fearful experiences and positive emotions linked to violent behaviour in the past. Additionally, visions for the future are developed in order to foster successful reintegration into society.

ELIGIBILITY:
Inclusion Criteria:

* Positive Emotions concerning aggressive behavior derived from expert interviews with higher Scores of the Appetitive Aggression Scale (AAS)
* children are part of an aid program for reintegration into society

Exclusion Criteria:

* current substance dependance or use of antipsychotic drugs
* chronically ill children

Ages: 12 Years to 23 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Positive emotions linked to aggressive behavior via the AAS-CS (Appetitive Aggressions Scale for children and students) | 6 months
Load of traumatic symptoms measured via the UCLA Adolescent PTSD Index (Clinician-administered PTSD scale) | 6 months

SECONDARY OUTCOMES:
Load of depressive symptoms measured via the MINI-KID | 6 months
Strength of suicidal ideation measured via the MINI-KID | 6 months
Functionality measured via the CGAS (Children's Global Assessment Scale) and SDQ (Strengths and Difficulties Questionnaire) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anselm Crombach, Dipl.-Psych., Principal Investigator — University of Constance
Locations (1):
- Fondation Stamm, Bujumbura, Bujumbura Mairie Province, Burundi